CLINICAL TRIAL: NCT01899612
Title: Vaginal Cytokines in Postmenopausal Women With Symptoms of Vulvovaginal Irritation
Brief Title: Vaginal Inflammation Markers in Postmenopausal Women With and Without Symptoms of Vaginal Inflammation
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 58/10
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Menopause; Vaginal Atrophy
Keywords: menopause; vaginal atrophy; cytokine; IL-1beta; IL-6; IL-8; TNF-alpha

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — vaginal lavage, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Symptomatic postmenopausal women: Postmenopausal women with vulvovaginal symptoms
- Asymptomatic postmenopausal women: Postmenopausal women without vulvovaginal symptoms

SUMMARY:
Many postmenopausal women suffer from vaginal symptoms such as dryness, itching, and painful intercourse. The underlying pathology is unknown. Since symptoms are comparable to those found in infectious vaginitis during the reproductive life stage, the investigators hypothesize that the vaginal milieu in symptomatic postmenopausal women is comparable to inflammation in vaginitis. The investigators therefore study vaginal cytokines in symptomatic and asymptomatic postmenopausal women.

DETAILED DESCRIPTION:
Background

Vulvovaginal irritation is a frequent complaint among postmenopausal women who are not on hormone therapy. Common symptoms include pruritus. Patients describe the irritation to be similar to that of vulvovaginal candidiasis during their reproductive years. Clinical improvement is seen with estrogen therapy. Most clinicians attribute the symptoms to vaginal dryness secondary to estrogen deficiency. However, the underlying pathophysiology of this clinical entity is not well defined. Since cytokines have been shown to play a significant role in the pathogenesis of infectious vaginitis, and there is evidence to suggest that estrogen influences cytokine production, we postulate that estrogen deficiency causes a disturbance in the vaginal cytokine environment similar to that of infectious vulvovaginitis.

Studies that investigate the pathogenesis of bacterial vaginosis, vulvovaginal candidiasis, and vestibulitis have identified changes in the level of antibodies and cytokines in the vagina during these processes. Donders and co-workers performed a study looking at the correlation between disturbance of the lactobacillary flora, vaginal pH, interleukin 1beta (IL-1b), and interleukin 8 (IL-8). Menopausal women were excluded from this study. Vaginal pH, IL-8, and IL-1β concentrations increased linearly with decreasing lactobacilli by 4 to 10 fold. IL-1β concentration was most closely related to decreasing lactobacilli, and IL-8 concentration was most closely related to positive culture results. Regúlez, Garcia Fernández, and co-worker performed a study to correlate the symptoms of vulvovaginal candidiasis with vaginal IgE levels. Patients who have clinically overt vulvovaginal candidiasis with classical symptomatology regardless of whether yeast or mycelia is identified in fresh smear or culture had higher IgE levels in their vagina than asymptomatic carriers or uninfected controls. This variation of host response has been proposed as one of the mechanism why only some women with vulvovaginal candidiasis experience symptoms. This concept of an imbalance between TH1 to TH2 cell reactivity with preference to the latter was further suggested by Puccetti, Romani and Bistoni. In contrary to the findings by Regúlez, Garcia Fernández and co-workers, Fidel, Ginsburg, and co-workers studied the vaginal-associated immunity in women with recurrent vulvovaginal candidiasis and found that Th-1 type response is increased. This area is certainly controversial and requires further investigations. Since IL-6 has been suggested as one of the cytokines involved in Th-2 or immediate-type hypersensitivity response, it will be of interest to study whether its level is increased for patients with symptomatology. Foster and Hasday compared the levels of IL-1b, and tumor necrosis factor-alpha (TNF-a) in perineal biopsy between women with vulvar vestibulitis and pain-free subjects, and found an increase in both cytokines in the former cases.

Estrogen has been shown to influence cytokine activity in the reproductive tract. García-Velasco and Arici published a review article on chemokines and human reproduction. In the article, the clinical relevance of chemokines in normal human reproductive events such as ovulation, menstruation, and implantation were summarized. There was however little information on their relevance in vaginal physiology. This is consistent with the little information on the topic of vaginal physiology in the literature. A study by Franklin, and Kutteh on the variation of immunoglobulins, and cytokines in cervical mucus in twelve women on oral contraceptives (OCs), and fifteen naturally cycling women showed a definite influence of exogenous and endogenous hormones on their levels. Cervical IgA, and IL-1b levels in women taking Ortho Novum 777® paralleled the increasing dosage of oral norethindrone, and the levels decreased after discontinuation of the oral contraceptive. Cervical IL-1b, and IL-10 both peaked just before ovulation in natural cycles. Cervical mucus IL-1b levels were found to correlate directly to changes in estrogen level during a natural cycle. Vaginal cytokine levels were not investigated in the study. Al-Harth, and co-workers measured cervicovaginal IL-1b, IL-4, IL-6, IL-8, IL-10, interferon-gamma (INF-gamma), transforming growth factor-beta (TGF-b), tumor necrosis factor-alpha (TNF-a), macrophage inflammatory protein-1alpha (MIP-1a) and TNG receptor II (TNFR II) during the follicular, and luteal phases of ovulatory cycle of six premenopausal women. Cervicovaginal IL-1b, and IL-6 were found to vary in level throughout the ovulatory cycle. Both IL-1b, and IL-6 were 5-fold higher in the follicular phase than in the luteal phase. Other cervicovaginal cytokines levels were not altered between the two phases. Plasma IL-8 level was higher in the follicular than luteal phase. The investigators' hypothesis is that postmenopausal estrogen deficiency causes changes in cytokine levels in the vagina similar to that found with vaginal candidiasis and bacterial vaginosis. A common cytokine etiology will account for the similarity of the symptomatology of infectious vaginitis and postmenopausal vaginal irritation.

Unpublished preliminary data from a study done on premenopausal women by Ballagh in the co-operating Howard and Georgeanna Jones Institute for Reproductive Medicine, Department of Obstetrics and Gynecology, Eastern Virginia Medical School, Norfolk, Virginia, USA, has shown that the mean levels of vaginal IL-1b and IL-8, as measured by ELISA, are higher in the luteal phase than the follicular phase in naturally cycling women. The median level of IL-1b is higher in the luteal phase than follicular phase but that of IL-8 is higher in the follicular phase than luteal phase. These results show that vaginal interleukin environment varies throughout the menstrual cycle to another. Women on oral contraceptive pills have increased mean levels of both vaginal IL-1b, and IL-8 compared to naturally cycling women. These data, though preliminary, support the theory that steroid hormone may play a role in the regulation of vaginal cytokine levels.

Objective

The principal goal of this pilot study is to determine the correlation between postmenopausal vulvovaginal irritative symptoms with vaginal interleukin levels. Cytokines to be evaluated in vaginal lavage will include IL-1β, IL-6, IL-8 and TNF-α. Plasma interleukin levels will be assessed concurrently, and compared to the vaginal levels to ensure that the vaginal levels obtained are not a result of contamination by plasma transudate. This study is thought to be the basis for a future randomised controlled trial involving the treatment of symptomatic menopausal women for investigation whether the resolution of the symptoms with e.g. estrogen and DHEA therapy is associated with a decrease in the interleukin levels.

Methods

Screening Investigations (visit 1):

History and physical examination Vaginal pH, KOH prep, whiff test, and wet prep for Trichomonas vaginalis Cervical sample for Neisseria gonorrhea & Chlamydia trachomatis assay

Enrollment Investigations (visit 2):

1. Vaginal pH
2. Vaginal smear for Nugent score and maturation index
3. Vaginal wet prep for Trichomonas vaginalis
4. Vaginal KOH prep and whiff test
5. Speculum examination and vaginal lavage
6. Leukocyte counts in vaginal samples
7. ELISA for serum IL-1b, IL-6, IL-8, TNF-a, IgE and estradiol
8. ELISA for IL-1b, IL-6, IL-8 TNF-a and IgE in vaginal lavage samples

ELIGIBILITY:
Inclusion Criteria:

* Age of 40 years or older
* At least 1 year history of amenorrhea
* Normal Pap smear within the past year
* Willingness to abstain from sexual intercourse and use of over-the-counter vaginal products for 7 days before the collection of vaginal samples
* Written informed consent.

Exclusion Criteria

* Administration of any form of oral hormone replacement therapy within 2 months, transdermal or vaginal hormone replacement therapy for 1 months prior to entry into the study
* Active vulvovaginal candidiasis, trichomonas vaginitis or bacterial vaginitis based on vaginal wet prep, pH, whiff test and KOH preparation;
* Untreated cervical, vaginal or vulvar intraepithelial neoplasia;
* Active sexually transmitted diseases including herpes simplex viral infection, gonorrhea and Chlamydia
* Pessary-users
* Active treatment with tamoxifen, raloxifene or other forms of selective estrogen receptor modulators (SERMs);
* Undiagnosed vaginal bleeding
* Hysterectomy
* Past or current history breast cancer, endometrial cancer or endometrial hyperplasia, hypertriglyceridemia or venous thromboembolism
* Immunocompromised patient including those with human immunodeficiency viral infection, chronic glucocorticoid use or active treatment with immunosuppressive agents

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects will be recruited at the menopause center, Inselspital Berne.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Difference in total vaginal IL-1beta in postmenopausal patients symptomatic, and asymptomatic of vulvovaginal irritation. | At enrolment (expected to be 2 weeks after screening)

SECONDARY OUTCOMES:
Difference in total vaginal IL-6 in postmenopausal patients symptomatic, and asymptomatic of vulvovaginal irritation. | At enrolment (expected to be 2 weeks after screening)
Difference in total vaginal IL-8 in postmenopausal patients symptomatic, and asymptomatic of vulvovaginal irritation. | At enrolment (expected to be 2 weeks after screening)
Difference in total vaginal TNF-alpha in postmenopausal patients symptomatic, and asymptomatic of vulvovaginal irritation. | At enrolment (expected to be 2 weeks after screening)
Difference in vaginal leukocyte counts in postmenopausal patients symptomatic, and asymptomatic of vulvovaginal irritation. | At enrolment (expected to be 2 weeks after screening)

CONTACTS AND LOCATIONS:
Overall Officials: Petra Stute, MD, Principal Investigator — Inselspital Bern Switzerland
Locations (1):
- Menopause Clinic, Women's Hospital, Inselspital Bern, Bern, Switzerland

REFERENCES:
- [Background] Notelovitz M, Mattox JH. Suppression of vasomotor and vulvovaginal symptoms with continuous oral 17beta-estradiol. Menopause. 2000 Sep-Oct;7(5):310-7. doi: 10.1097/00042192-200007050-00005. PMID 10993030
- [Background] Al-Harthi L, Wright DJ, Anderson D, Cohen M, Matity Ahu D, Cohn J, Cu-Unvin S, Burns D, Reichelderfer P, Lewis S, Beckner S, Kovacs A, Landay A. The impact of the ovulatory cycle on cytokine production: evaluation of systemic, cervicovaginal, and salivary compartments. J Interferon Cytokine Res. 2000 Aug;20(8):719-24. doi: 10.1089/10799900050116426. PMID 10954915
- [Background] Franklin RD, Kutteh WH. Characterization of immunoglobulins and cytokines in human cervical mucus: influence of exogenous and endogenous hormones. J Reprod Immunol. 1999 Mar;42(2):93-106. doi: 10.1016/s0165-0378(98)00086-2. PMID 10221733
- [Derived] Kollmann Z, Bersinger N, von Wolff M, Thurman AR, Archer DF, Stute P. Vaginal cytokines do not correlate with postmenopausal vulvovaginal symptoms. Gynecol Endocrinol. 2015 Apr;31(4):317-21. doi: 10.3109/09513590.2014.995080. Epub 2015 Jan 5. PMID 25559048